CLINICAL TRIAL: NCT03474341
Title: Preoperative Image-guided Identification of Response to Neoadjuvant Chemoradiotherapy in Esophageal Cancer
Acronym: PRIDE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: University Medical Center Groningen (Other); The Netherlands Cancer Institute (Other); Koningin Wilhelmina Fonds (Other); Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Gert Meijer, PhD, Clinical Physicist at the Department of Radiation Oncology, UMC Utrecht
Other Study IDs: NL62881.041.17; Project ID 10291 (Other Grant/Funding Number: Koningin Wilhelmina Fonds (KWF) Kankerbestrijding); 17-941 (Other: Medical Ethical Committee UMC Utrecht)
Record Dates: First submitted 2018-01-30; First posted 2018-03-22 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Esophageal Cancer; Esophageal Adenocarcinoma; Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms
Keywords: Neoadjuvant chemoradiotherapy (nCRT); Pathologic complete response (pCR); Magnetic Resonance Imaging (MRI); PET-CT; Circulating tumor DNA (ctDNA); endoscopy
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma; Pathologic Complete Response | interventions — Magnetic Resonance Imaging; Diffusion Magnetic Resonance Imaging; Dynamic Contrast Enhanced Magnetic Resonance Imaging; Positron Emission Tomography Computed Tomography; Endoscopy; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Resectable esophageal squamous cell- or adenocarcinoma: Patients (>18 years) with potentially resectable locally advanced squamous cell- or adenocarcinoma of the esophagus or gastroesophageal junction, receiving nCRT according to the CROSS regimen prior to surgery.
  CROSS regimen: weekly carboplatin (doses titrated to achieve an area under the curve of 2 mg per milliliter per minute) and paclitaxel (50 mg per square meter of body-surface area) for 5 weeks and concurrent radiotherapy (41.4 Gy in 23 fractions, delivered 5 days per week on workdays with intensity modulated radiotherapy, including photon and proton therapy)
  Interventions: Diagnostic Test: MRI; Diagnostic Test: PET-CT; Diagnostic Test: Endoscopy; Diagnostic Test: Blood samples

INTERVENTIONS:
Diagnostic Test: MRI — * Anatomical (T2W) and functional MRI (DWI and DCE) at a 1.5T Siemens or Philips scanner
  * DWI series: sagittal (sIVIM) and high-resolution transversal (HR tDWI)
  * DCE serie: dynamic20
  * In total, three MRI scan series (before, during, after nCRT)
  * Measurements: i.a. change in apparent diffusion coefficient (ADC) or area-under-the-gadolinium-concentration time curve (AUC) within tumor delineation over time, radiological (qualitative) assessment of residual disease
  Other Names: Magnetic Resonance Imaging; DW-MRI; DCE-MRI; T2W
Diagnostic Test: PET-CT — * According to European Association of Nuclear Medicine (EANM) Research Ltd guidelines (EARL)
  * In total one additional PET-CT (during nCRT) for study purposes. A PET-CT scan at diagnosis and after nCRT are included in the standard diagnostic work-up for esophageal cancer.
  * Measurements: i.a. change in TLG (Total Lesion Glycolysis), SUVmax (Standardized Uptake Value) or Ktrans within tumor delineation over time
  Other Names: 18-F FDG PET-CT; PET
Diagnostic Test: Endoscopy — Additional endoscopy and/or endoscopic ultrasonography (EUS) with biopsies of the primary tumor site and other suspected lesions in the esophagus after completion of nCRT and prior to surgery
  Other Names: Endoscopic assessment; EUS
Diagnostic Test: Blood samples — * Blood samples at three different time points (before, during and after nCRT) will be collected
  * Blood will be collected in cell-free DNA collection tubes
  * Purpose: isolation of ctDNA and subsequent mutation analysis by means of Next Generation Sequencing
  * Measurements: the presence of, and changes in, ctDNA during nCRT
  Other Names: ctDNA

SUMMARY:
Rationale: For locally advanced esophageal cancer the standard treatment consists of 5 weeks of neoadjuvant chemoradiotherapy (nCRT) followed by surgery. Surgery is currently performed independent of the response to nCRT and is associated with substantial morbidity. Prior knowledge of the eventual response to nCRT would greatly impact on the optimal care for many esophageal cancer patients for two imperative reasons:

Firstly, it is argued that patients who achieved a pathologic complete response (pCR, 29%) may not have benefitted from surgery. Consequently, proper identification of pathological complete responders prior to surgery could yield an organ-preserving regimen avoiding unnecessary toxicity.

Secondly, non-responders are exposed to the side effects of nCRT without showing any tumor regression. Early identification of the non-responders during nCRT would be beneficial for this group as ineffective therapy could be stopped, and for who altered treatment strategies could be explored.

Objective: To develop a multimodal model that predicts the probability of pathologic complete response to nCRT in esophageal cancer, by integrating diffusion weighted magnetic resonance imaging (DW-MRI) and dynamic contrast enhanced magnetic resonance imaging (DCE-MRI) in conjunction with combined 18F-fluorodeoxyglucose positron emission tomography and computed tomography (18F-FDG PET-CT) scans acquired prior to, during and after administration of nCRT.

Study design: Multi-center observational study

Study population: Patients (>18 years) with potentially resectable locally advanced squamous cell- or adenocarcinoma of the esophagus or gastroesophageal junction, receiving nCRT prior to surgery.

Intervention: In addition to the standard diagnostic work-up for esophageal cancer that includes a 18F-FDG PET-CT scan at diagnosis and after nCRT, one 18F-FDG PET-CT scans will be performed during nCRT, as well as three MRI scans (before, during and after nCRT) within fixed time intervals. Furthermore, after response imaging after nCRT has been performed, but prior to surgery, patients will undergo (on an opt-out basis) an endoscopy and/or endoscopic ultrasonography (EUS) with biopsies of the primary tumor site, other suspected lesions and suspected lymph nodes. Furthermore, blood samples will be collected at three time points.

Main study parameters/endpoints: An accurate multimodal prediction model for the patients' individual probability of pathologic complete response after nCRT, based on the quantitative parameters derived from a longitudinal series of DW-MRI, DCE-MRI and 18F-FDG PET-CT datasets.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma or adenocarcinoma of the esophagus or gastroesophageal junction (i.e. tumors involving both cardia and esophagus on endoscopy)
* Potentially resectable locally advanced esophageal tumor (cT1b-4a N0-3 M0): based on standard primary staging by EUS and 18F-FDG PET-CT
* Scheduled to receive neoadjuvant chemoradiotherapy according to CROSS-regimen1: weekly administration of carboplatin and paclitaxel for 5 weeks and concurrent radiotherapy (41.4 Gray in 23 fractions, 5 days per week) followed by esophagectomy
* Age > 18 years

Exclusion Criteria:

* Patients who meet exclusion criteria for MRI
* Patients who meet exclusion criteria for intravenous gadolinium-based contrast:

  * Glomerular Filtration Rate (GFR) of <30 mL/min/1.73m2
  * Nephrogenic Systemic Fibrosis (strict contra-indication for gadolinium-based contrast)
  * Known allergy for gadolinium-based contrast
* Patients with a blood plasma glucose concentration >10 mmol/L or poorly controlled diabetes mellitus
* Endoscopic mucosal resection (EMR) or endoscopic submucosal dissection (ESD) of primary tumor prior to start of neoadjuvant chemoradiotherapy
* Pregnant or breast-feeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with resectable esophageal or gastroesophageal junction adeno- or squamous cell carcinoma, scheduled to receive neoadjuvant chemoradiotherapy according to the CROSS-regimen
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-04-09 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Histopathologic response | Based on resection specimen (surgery 8-10 weeks after finishing nCRT)
  Histopathologic response of the primary tumor to nCRT according to the tumor regression grade (TRG) scale as determined by expert pathologist.
  TRG 1: no residual viable tumor cells, pathologic complete response TRG 2: rare residual cancer cells TRG 3: predominant fibrosis with increased number of residual cancer cells TRG 4: residual cancer outgrowing fibrosis or no regressive change

SECONDARY OUTCOMES:
Pathological T- and N-stage | Based on resection specimen (surgery 8-10 weeks after finishing nCRT)
  Pathological T- and N-stage as determined by expert pathologist (based on the American Joint Committee on Cancer [AJCC] Tumor Node Metastasis [TNM] staging system)
Disease-free survival. | Up to 5-year follow-up
  Disease-free survival based on local follow-up policies (time to locoregional or distal recurrence of esophageal cancer).
Overall survival. | Up to 5-year follow-up
  Overall survival based on local follow-up policies.

CONTACTS AND LOCATIONS:
Overall Officials: Gert J Meijer, PhD, Principal Investigator — UMC Utrecht; Marcel Verheij, MD, PhD, Principal Investigator — Antoni van Leeuwenhoek - Netherlands Cancer Institute; J. (Hans) A. Langendijk, MD, PhD, Principal Investigator — University Medical Center Groningen; Hanneke WM van Laarhoven, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (4):
- Netherlands (4):
  - Amsterdam University Medical Centers, Academic Medical Center, Amsterdam
  - Antoni van Leeuwenhoek - Netherlands Cancer Institute (NKI-AVL), Amsterdam
  - University Medical Center Groningen (UMCG), Groningen
  - University Medical Center Utrecht (UMCU), Utrecht

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Borggreve AS, Mook S, Verheij M, Mul VEM, Bergman JJ, Bartels-Rutten A, Ter Beek LC, Beets-Tan RGH, Bennink RJ, van Berge Henegouwen MI, Brosens LAA, Defize IL, van Dieren JM, Dijkstra H, van Hillegersberg R, Hulshof MC, van Laarhoven HWM, Lam MGEH, van Lier ALHMW, Muijs CT, Nagengast WB, Nederveen AJ, Noordzij W, Plukker JTM, van Rossum PSN, Ruurda JP, van Sandick JW, Weusten BLAM, Voncken FEM, Yakar D, Meijer GJ; PRIDE study group. Preoperative image-guided identification of response to neoadjuvant chemoradiotherapy in esophageal cancer (PRIDE): a multicenter observational study. BMC Cancer. 2018 Oct 20;18(1):1006. doi: 10.1186/s12885-018-4892-6. PMID 30342494